CLINICAL TRIAL: NCT05846633
Title: Effectiveness of C-Mill Treadmill Training Versus Conventional Treadmill on Balance and Psychological Status in Elderly Population: A Randomized Clinical Trial
Brief Title: Effectiveness of C-Mill Treadmill Training Versus Conventional Treadmill on Balance and Psychological Status in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Ayman Mohammed Zafer, PhD Candidate in neurological rehabilitation Sciences, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-PGS-2023-03-253
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Elderly; Geriatric
Keywords: elderly; fall risk; gait; balance; virtual reality; treadmill

STUDY DESIGN:
Who Masked: Participant
Masking Description: the participants will be randomly assigned to 2 groups for intervention, none of them knows which arm will be for intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR treadmill (Experimental): The intervention of this study will be C-Mill virtual reality treadmill (Motekforce Link, Amsterdam/Culemborg, The Netherlands).
  Sixteen participants will be included in the c-mill treadmill program for 50 minutes per session / two sessions per week, over six successive weeks (a total of 12 sessions).
  Every participant will be trained for (50 minutes) as follows: warming up by walking on the treadmill with a comfortable walking speed upon individual's capability for 5 minutes. The speed should be determined for each one. Then participants continue training on the treadmill for 20 minutes. Visually guided stepping exercises will be applied. Participants should get a (5-min break) and then resume training on the treadmill for 25 minutes. Obstacle avoidance exercises and Walking area practice will be applied.
  Interventions: Device: C mell treadmill
- Conventional group (Active Comparator): Like group I, each participant will be trained on a conventional treadmill for (50 minutes) as follows: warming up by walking on the treadmill belt with a comfortable walking speed suitable for each participant for 5 minutes. The speed should be determined Then participants continue training on the treadmill for 20 minutes; no VR will be used or applied. Participants should get a 5-min break and then resume training on the treadmill again for 25 minutes.
  Interventions: Device: C mell treadmill

INTERVENTIONS:
Device: C mell treadmill — C Mell treadmill provides Virtual Reality environment for rehabilitation with obstacles and motivational assistance

SUMMARY:
Background: Aging is characterized by reduced cognitive and physical functions; consequently, balance, falling and different activities of daily living get exaggerated reductions. Psychological status and falling are related bidirectionally. Depression is a common mental or mood disorder affecting more than 264 million people worldwide. It is a recurrent state of unhappiness and loss of interest. It is not simple as fluctuating mood because of short emotional response. To prevent falling, functional mobility and impairment of balance should be addressed. Many studies have shown that treadmill training is effective in improving the elderly person's ability to walk. The C-Mill treadmill afford a safe virtual reality environment and challenging obstacles and balance games, which increase of walking and improve everyday life performance. Aims: This study aims are to investigate the clinical effectiveness of virtual reality treadmill training on psychological status and balance in elderly population in addition to compare the significant differences between them. Materials & Methods: Fifty-Eight elderly participants will be equally and randomly assigned to Group-I: Twenty-Nine participants will be trained on C-Mill treadmill for 50 minutes per session /2 session /week for six successive weeks. Group-II: Twenty-Nine participants will be trained on conventional treadmill for 50 minutes per session /2 session /week for six successive weeks. Psychological status and Depression will be evaluated by using the Depression Anxiety Stress Scale-2, Geriatric Depression Scale and the Beck Depression Inventory while the balance will be evaluated by using Berge balance scale and timed up and go test, whereas the functional capacity will be measured by using 6 MWT. Statistical analysis: The data will be statistically analysis by using (SPSS version 25). The Shapiro walk test will be used to examine the normality of data distribution. Independent t- test will be used to determine significant differences between two groups (between groups) and paired t- test to determine significant differences before and after intervention in both groups. Significance level at <0.05 and confidence interval CI with 95%.

DETAILED DESCRIPTION:
Fifty-Eight elderly participants will be equally and randomly assigned to Group-I: Twenty-Nine participants will be trained on C-Mill treadmill for 50 minutes per session /2 session /week for six successive weeks. Group-II: Twenty-Nine participants will be trained on conventional treadmill for 50 minutes per session /2 session /week for six successive weeks. Psychological status and Depression will be evaluated by using the Depression Anxiety Stress Scale-2, Geriatric Depression Scale and the Beck Depression Inventory while the balance will be evaluated by using Berge balance scale and timed up and go test, whereas the functional capacity will be measured by using 6 MWT

ELIGIBILITY:
Inclusion Criteria:

* elderly male & female (60-75 years old) subjects will participate in this study. Based on a confirmed written medical report and signed by their physicians. They should be with controlled and stable medical condition, neither Vit-D deficient nor thyroid affected. Participants should have an acceptable level of cognitive function (score 25 or more on Mini-Mental State Examination, score 40 or less on Berg Balance Scale (BBSand score more than 5 on Geriatric Depression Scale (GDS).

All participants should not receive other training to improve their balance and gait other than the protocol of this study.

Exclusion Criteria:

Participants will be excluded if they have one of the following conditions:

* Medically unstable
* Fxed lower limb bony deformities
* Muscle paralysis,
* Cerebellar impairment,
* Visual problems,
* Vestibular problems,
* Cognitive reduction, any condition may lead to problematic exercises
* Using vertigo or anti-seizures medications,
* Score more than 40 on Berg Balance Scale (BBS)
* Score less than 5 on Geriatric Depression Scale (GDS).

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-05-02 (Estimated); Study Completion 2024-05-02 (Estimated)

PRIMARY OUTCOMES:
Biodex Balance System (BBS; Biodex Inc., Shirley, NY) | 6 Weeks
  It will be utilized as a reliable and valid device for measuring balance stability during standing in both static and dynamic situations (Cachupe et al.,2001 and Chen et al., 2014). Two balance tests will be performed: Limit of Stability (LOS) and Fall risk test. Both tests challenge the ability of participants to control and maintain balance by maintaining their center of gravity within their base of support. The Biodex system has both a static and dynamic mode with 12 levels of platform tilt (greatest stability level = level 12; least stability level = level 1). The static mode and dynamic level (11) of platform tilt will be e selected in this study to perform PST and LOS tests.
Berg Balance Scale | 6 weeks
  a 14-item list; each will be scored ranging from (0-4); 0 is the lowest and 4 is the highest function (0 -20 = high fall risk, 21-40 = medium fall risk and 41-56 = low fall risk). This tool is valid and reliable
The Timed Up and Go Test (TUG) | 6 weeks
  It will be used to assess the following parameters in older adults: fall risk, walking ability, balance, and mobility. Participants while wearing regular footwear will start from sitting position by standing up upon therapist's command; walk forward for 3 meters, turn around, walk back to the chair and sit down when timing should stop. Any assistive devices should be noted. It is a reliable, valid, and sensitive test that is a specific measure of the probability for falls among elderly.
The six-minute walk test (6MWT) | 6 Weeks
  It will assess the distance that the participant's walking capacity for a total of six minutes on a hard, uneven surface. The 6MWT was originally developed in frail elderly patients aged 60-90 years referred to a geriatric hospital. It has been used to determine exercise tolerance changes following interventions for healthy older adults
The Beck Depression Inventory (BDI) | 6 Weeks
  It is a 21-items and self-report form used to assess the presence and severity of symptoms of depression in adults (13-80 years old). Questions should be answered upon participant's feeling during last 2 weeks. The BDI takes approximately 10 minutes to complete. The higher the Beck score the higher the feelings of depression; (1-10) These ups and downs are considered normal, (11-16) mild mood disturbance (17-20) borderline clinical depression (21-30) moderate depression (31-40) severe depression above 40 reflects extreme depression. This tool is reliable and has been validated and standardized on geriatric population with relatively less somatic-related items
Geriatric Depression Scale - 15 (short form) (GDS-15) | 6 Weeks
  It is a 15-items, and self-report form. All are YES/NO question, each is worth one point and should be answered based on participant's feeling over last week. 10 items indicate presence of depression if answered positively, while the other 5 indicate depression if answered negatively. This form can be completed in approximately 5 to 7 minutes. This tool has been validated and has a high correlation with depressive symptoms and differentiates between depressed from non-depressed patients. It is valid and reliable scale in geriatrics with a cut-off score of 6 on GDS-15 has 94% sensitivity and 85% specificity in community dwelling older adults, while a cut-off score of 5 has 72% sensitivity and 78% specificity in home care patients
Depression in Old Age Scale (DIA-S | 6 Weeks
  is a self-report instrument consists of ten (Yes/No) short statements that focus on emotional, motivational, and cognitive symptoms of . It has a higher specificity and internal consistency (Heidenblut & Zank, 2010). This tool is recommended for research and clinical practice (Heidenblut & Zank, 2020). Score ranges from (0-10); where (0 = no depressive symptoms) and (10 = maximal depressive symptoms); where 4 is an indicative for a depressive disorder.
Depression Anxiety Stress Scale-21 (DASS-21) Arabic version | 6 Weeks
  is a self-report instrument that consists of three domains; each domain has seven items. Using a four-point Likert scale (0-3), it assesses the negative emotional symptoms. 3 indicates higher severity of negative symptoms. The three domains are: Depression scale, Anxiety scale, and Stress scale. This tool is valid and has excellent reliability.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alabdullgader A, Rabbani U. Prevalence and Risk Factors of Falls Among the Elderly in Unaizah City, Saudi Arabia. Sultan Qaboos Univ Med J. 2021 Feb;21(1):e86-e93. doi: 10.18295/squmj.2021.21.01.012. Epub 2021 Mar 15. PMID 33777428
- [Background] Alghnam S, Alsayyari AS, Towhari JA, Alsayer RM, Almohaimeed MY, Aldebasi MH, Albabtin IT. Epidemiological characteristics of fall injuries and their related outcome in Riyadh, Saudi Arabia: A descriptive study from a Level-I trauma center. J Family Community Med. 2020 May-Aug;27(2):114-119. doi: 10.4103/jfcm.JFCM_245_19. Epub 2020 Jun 3. PMID 32831557
- [Background] Ali AM, Ahmed A, Sharaf A, Kawakami N, Abdeldayem SM, Green J. The Arabic Version of The Depression Anxiety Stress Scale-21: Cumulative scaling and discriminant-validation testing. Asian J Psychiatr. 2017 Dec;30:56-58. doi: 10.1016/j.ajp.2017.07.018. Epub 2017 Jul 18. PMID 28755630
- [Background] Almegbel FY, Alotaibi IM, Alhusain FA, Masuadi EM, Al Sulami SL, Aloushan AF, Almuqbil BI. Period prevalence, risk factors and consequent injuries of falling among the Saudi elderly living in Riyadh, Saudi Arabia: a cross-sectional study. BMJ Open. 2018 Jan 10;8(1):e019063. doi: 10.1136/bmjopen-2017-019063. PMID 29326189
- [Background] Alshammari SA, Alhassan AM, Aldawsari MA, Bazuhair FO, Alotaibi FK, Aldakhil AA, Abdulfattah FW. Falls among elderly and its relation with their health problems and surrounding environmental factors in Riyadh. J Family Community Med. 2018 Jan-Apr;25(1):29-34. doi: 10.4103/jfcm.JFCM_48_17. PMID 29386959
- [Background] Ashworth NL, Chad KE, Harrison EL, Reeder BA, Marshall SC. Home versus center based physical activity programs in older adults. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD004017. doi: 10.1002/14651858.CD004017.pub2. PMID 15674925
- [Background] Beck, A. T., Steer, R. A., & Carbin, M. G. (1988). Psychometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clinical psychology review, 8(1), 77-100.
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Berger-Vachon, C. (2006). Virtual reality and disability. Technology and Disability, 18(4), 163-165.
- [Background] Berry, B. D. (2013). Effects of upper body resistance while treadmill walking in older adults (Doctoral dissertation, Wichita State University).
- [Background] Blazer DG. Depression in late life: review and commentary. J Gerontol A Biol Sci Med Sci. 2003 Mar;58(3):249-65. doi: 10.1093/gerona/58.3.m249. PMID 12634292
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Britton A, Shipley M, Singh-Manoux A, Marmot MG. Successful aging: the contribution of early-life and midlife risk factors. J Am Geriatr Soc. 2008 Jun;56(6):1098-105. doi: 10.1111/j.1532-5415.2008.01740.x. Epub 2008 May 12. PMID 18482302
- [Background] Burns ER, Stevens JA, Lee R. The direct costs of fatal and non-fatal falls among older adults - United States. J Safety Res. 2016 Sep;58:99-103. doi: 10.1016/j.jsr.2016.05.001. Epub 2016 May 28. PMID 27620939
- [Background] Cabeza, R., Nyberg, L., & Park, D. C. (Eds.). (2016). Cognitive neuroscience of aging: Linking cognitive and cerebral aging. Oxford University Press.
- [Background] Cachupe, W. J., Shifflett, B., Kahanov, L., & Wughalter, E. H. (2001). Reliability of biodex balance system measures. Measurement in physical education and exercise science, 5(2), 97-108.
- [Background] Cakit BD, Saracoglu M, Genc H, Erdem HR, Inan L. The effects of incremental speed-dependent treadmill training on postural instability and fear of falling in Parkinson's disease. Clin Rehabil. 2007 Aug;21(8):698-705. doi: 10.1177/0269215507077269. PMID 17846069
- [Background] Cesari M, Landi F, Torre S, Onder G, Lattanzio F, Bernabei R. Prevalence and risk factors for falls in an older community-dwelling population. J Gerontol A Biol Sci Med Sci. 2002 Nov;57(11):M722-6. doi: 10.1093/gerona/57.11.m722. PMID 12403800
- [Background] Chand SP, Arif H, Kutlenios RM. Depression (Nursing). 2023 Jul 17. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK568733/ PMID 33760492
- [Background] Chen CH, Lin SF, Yu WH, Lin JH, Chen HL, Hsieh CL. Comparison of the test-retest reliability of the balance computerized adaptive test and a computerized posturography instrument in patients with stroke. Arch Phys Med Rehabil. 2014 Aug;95(8):1477-83. doi: 10.1016/j.apmr.2014.03.005. Epub 2014 Mar 21. PMID 24662809
- [Background] Cho GH, Hwangbo G, Shin HS. The Effects of Virtual Reality-based Balance Training on Balance of the Elderly. J Phys Ther Sci. 2014 Apr;26(4):615-7. doi: 10.1589/jpts.26.615. Epub 2014 Apr 23. PMID 24764645
- [Background] Cobb, S., Brooks, T., Sharkey, P. M., & Merrick, J. (2006). Virtual reality and disability [Editorial]. International Journal on Disability and Human Development, 5(2), 95-96. https://doi.org/10.1515/IJDHD.2006.5.2.95
- [Background] Crosbie JH, Lennon S, Basford JR, McDonough SM. Virtual reality in stroke rehabilitation: still more virtual than real. Disabil Rehabil. 2007 Jul 30;29(14):1139-46; discussion 1147-52. doi: 10.1080/09638280600960909. PMID 17613000
- [Background] Cuijpers P, van Straten A, Smit F. Psychological treatment of late-life depression: a meta-analysis of randomized controlled trials. Int J Geriatr Psychiatry. 2006 Dec;21(12):1139-49. doi: 10.1002/gps.1620. PMID 16955421
- [Background] de Rooij, I. J., van de Port, I. G., & Meijer, J. W. G. (2017). Feasibility and effectiveness of virtual reality training on balance and gait recovery early after stroke: a pilot study. Walking in relation to participation after stroke, 129.
- [Background] Deandrea S, Lucenteforte E, Bravi F, Foschi R, La Vecchia C, Negri E. Risk factors for falls in community-dwelling older people: a systematic review and meta-analysis. Epidemiology. 2010 Sep;21(5):658-68. doi: 10.1097/EDE.0b013e3181e89905. PMID 20585256
- [Background] Deshpande N, Metter EJ, Lauretani F, Bandinelli S, Guralnik J, Ferrucci L. Activity restriction induced by fear of falling and objective and subjective measures of physical function: a prospective cohort study. J Am Geriatr Soc. 2008 Apr;56(4):615-20. doi: 10.1111/j.1532-5415.2007.01639.x. Epub 2008 Feb 26. PMID 18312314
- [Background] Dockx K, Bekkers EM, Van den Bergh V, Ginis P, Rochester L, Hausdorff JM, Mirelman A, Nieuwboer A. Virtual reality for rehabilitation in Parkinson's disease. Cochrane Database Syst Rev. 2016 Dec 21;12(12):CD010760. doi: 10.1002/14651858.CD010760.pub2. PMID 28000926
- [Background] Dusemund F, Steiner M, Vuilliomenet A, Muller C, Bossart R, Regez K, Schild U, Conca A, Huber A, Reutlinger B, Muller B, Albrich WC. Multidisciplinary Assessment to Personalize Length of Stay in Acute Decompensated Heart Failure (OPTIMA II ADHF). J Clin Med Res. 2012 Dec;4(6):402-9. doi: 10.4021/jocmr1154w. Epub 2012 Nov 11. PMID 23226173
- [Background] Fokkenrood HJ, Bendermacher BL, Lauret GJ, Willigendael EM, Prins MH, Teijink JA. Supervised exercise therapy versus non-supervised exercise therapy for intermittent claudication. Cochrane Database Syst Rev. 2013 Aug 23;(8):CD005263. doi: 10.1002/14651858.CD005263.pub3. PMID 23970372
- [Background] Galea M, Woodward M. Mini-Mental State Examination (MMSE). Aust J Physiother. 2005;51(3):198. doi: 10.1016/s0004-9514(05)70034-9. No abstract available. PMID 16187459
- [Background] Gao Z, Lee JE, McDonough DJ, Albers C. Virtual Reality Exercise as a Coping Strategy for Health and Wellness Promotion in Older Adults during the COVID-19 Pandemic. J Clin Med. 2020 Jun 25;9(6):1986. doi: 10.3390/jcm9061986. PMID 32630367
- [Background] Gaugler JE, Reese M, Mittelman MS. Effects of the Minnesota Adaptation of the NYU Caregiver Intervention on Depressive Symptoms and Quality of Life for Adult Child Caregivers of Persons with Dementia. Am J Geriatr Psychiatry. 2015 Nov;23(11):1179-92. doi: 10.1016/j.jagp.2015.06.007. Epub 2015 Jun 25. PMID 26238226
- [Background] Goble DJ, Cone BL, Fling BW. Using the Wii Fit as a tool for balance assessment and neurorehabilitation: the first half decade of "Wii-search". J Neuroeng Rehabil. 2014 Feb 8;11:12. doi: 10.1186/1743-0003-11-12. PMID 24507245
- [Background] Grabiner MD, Kaufman KR. Developing and Establishing Biomechanical Variables as Risk Biomarkers for Preventable Gait-Related Falls and Assessment of Intervention Effectiveness. Front Sports Act Living. 2021 Sep 22;3:722363. doi: 10.3389/fspor.2021.722363. eCollection 2021. PMID 34632378
- [Background] Groth-Marnat, G. (2009). Handbook of psychological assessment. John Wiley & Sons.
- [Background] Haddad M. Depression in adults with a chronic physical health problem: treatment and management. Int J Nurs Stud. 2009 Nov;46(11):1411-4. doi: 10.1016/j.ijnurstu.2009.08.007. No abstract available. PMID 19748379
- [Background] Harada ND, Chiu V, Stewart AL. Mobility-related function in older adults: assessment with a 6-minute walk test. Arch Phys Med Rehabil. 1999 Jul;80(7):837-41. doi: 10.1016/s0003-9993(99)90236-8. PMID 10414771
- [Background] Heidenblut S, Zank S. Screening for Depression in Old Age With Very Short Instruments: The DIA-S4 Compared to the GDS5 and GDS4. Gerontol Geriatr Med. 2020 Dec 10;6:2333721420981328. doi: 10.1177/2333721420981328. eCollection 2020 Jan-Dec. PMID 33354593
- [Background] Heinzel, S., Lawrence, J. B., Kallies, G., Rapp, M. A., & Heissel, A. (2015). Using exercise to fight depression in older adults: A systematic review and meta-analysis. GeroPsych: The Journal of Gerontopsychology and Geriatric Psychiatry, 28(4), 149.
- [Background] Hu S, Tucker L, Wu C, Yang L. Beneficial Effects of Exercise on Depression and Anxiety During the Covid-19 Pandemic: A Narrative Review. Front Psychiatry. 2020 Nov 4;11:587557. doi: 10.3389/fpsyt.2020.587557. eCollection 2020. PMID 33329133
- [Background] Iaboni A, Flint AJ. The complex interplay of depression and falls in older adults: a clinical review. Am J Geriatr Psychiatry. 2013 May;21(5):484-92. doi: 10.1016/j.jagp.2013.01.008. Epub 2013 Feb 6. PMID 23570891